CLINICAL TRIAL: NCT02504983
Title: Randomized, Open Label, Clinical Trial for GALNT14 Genotype - Guided, Sorafenib in Combination With TACE Therapy in Hepatocellular Carcinoma
Brief Title: Clinical Trial for GALNT14 Genotype - Guided, Sorafenib in Combination With TACE in Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104-1686A3
Record Dates: First submitted 2015-07-16; First posted 2015-07-22 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: SNPs
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GALNT14 TT (Active Comparator): Patients will be treated by Transcatheter arterial chemoembolization every 12 ± 2 weeks dependent on CT evaluation. Before each TACE, dynamic CT will be performed for pre-treatment evaluation. When no viable tumor is seen on CT, TACE is to be discontinued.
  Interventions: Procedure: TACE
- GALNT14 non-TT TACE alone (Active Comparator): Patients will be treated by Transcatheter arterial chemoembolization every 12 ± 2 weeks dependent on CT evaluation. Before each TACE, dynamic CT will be performed for pre-treatment evaluation. When no viable tumor is seen on CT, TACE is to be discontinued.
  Interventions: Procedure: TACE
- GALNT14 non-TT TACE plus sorafenib (Experimental): Patients will be treated by Transcatheter arterial chemoembolization every 12 ± 2 weeks dependent on CT evaluation, plus sorafenib adjuvant therapy. Before each TACE, dynamic CT will be performed for pre-treatment evaluation. When no viable tumor is seen on CT, TACE is to be discontinued. patients will receive sorafenib 400 mg/d between each TACE. Patient will start receiving Sorafenib on Day 4 (up to Day 7) after 1st TACE (Day 1) and will interrupt after evening dose 4 days before each next TACE and re-start Sorafenib on Day 4 (up to Day 7) after each TACE cycle.Additional sorafenib treatment is optional and will be judged by investigator in the subject's best medical interest.
  Interventions: Drug: sorafenib; Procedure: TACE

INTERVENTIONS:
Drug: sorafenib — sorafenib is an oral, multikinase inhibitor approved for the treatment of advanced hepatocellular carcinoma
  Other Names: Nexavar
  Arms: GALNT14 non-TT TACE plus sorafenib
Procedure: TACE — Transcatheter arterial chemoembolization was performed by the injection of small embolic particles coated with chemotherapeutic agents selectively into an artery directly supplying a tumor.
  Other Names: Transcatheter arterial chemoembolization

SUMMARY:
Transcatheter arterial chemoembolization (TACE) + sorafenib therapy has been demonstrated to exert a beneficial effective on time-to-tumor-progression (TTP) in patients with unresectable hepatocellular carcinoma (HCC) in some studies. However, the beneficial effect varies among studies conducted in different areas of the world. The objectives of this study are (1) to understand whether GALNT14 TT genotype patients respond better than do GALNT14 non-TT genotype patients when treated by TACE; and (2) to understand whether GALNT14 non-TT genotype patients can benefit from TACE plus sorafenib (Nexavar) combination therapy. Patients enrolled will be stratified by GALNT14 genotyping. The GALNT14 "non-TT" patients were then randomized into two subgroups to evaluate the safety, tolerability and efficacy of TACE plus sorafenib therapy.

The primary endpoint of this study is the efficacy of TACE with or without sorafenib combination therapy evaluated by complete remission (CR).

The secondary endpoints are:

1. Time to partial or complete response (PR + CR).
2. Time-to-tumor-progression (TTP) and the progression free survival (PFS).
3. Overall survival (OS).
4. Safety and tolerability of TACE plus sorafenib therapy.

DETAILED DESCRIPTION:
The strategy of TACE + sorafenib is now being intensively investigated. It is a safe approach with significant beneficial effect on TTP in some studies, but the beneficial effect on OS remains uncertain. In the present study, we hypothesized that the GALNT14 genotype might play a role in this issue. Our pilot study indicated that GALNT14 "TT" genotype was associated with a favorable complete response rate in patients treated by TACE alone. This genotype was present in ~ 25% of Chinese population coming from Taiwan, Colorado (US), or Beijing (China), and in ~ 7% of Italian population. But it was present in ~ 50% of Japanese population. The lower percentage of a TACE - favorable genotype in Chinese and Italian population could explain the different results between Japanese and Chinese/Italian clinical trials. It is possible that in a population with higher percentage of TACE - favorable genotype (GALNT14 "TT"), the beneficial effect of sorafenib adjuvant treatment might not be detected. In this study, we proposed to examine the TACE + sorafenib effect in patients with GALNT14 "non-TT" genotype, a TACE - unfavorable genotype.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed Diagnosis of HCC:

   Cirrhotic subjects: Clinical diagnosis by AASLD criteria HCC can be defined in cirrhotic subjects by one imaging technique (CT scan, MRI, or second generation contrast ultrasound) showing a nodule larger than 2cm with contrast uptake in the arterial phase and washout in venous or late phases, or two imaging techniques showing this radiological behaviour for nodules of 1-2cm in diameter Cytohistological confirmation is required for subjects who do not fulfill these eligibility criteria

   Non-cirrhotic subjects:

   For subjects without cirrhosis, histological confirmation is mandatory Documentation of original biopsy for diagnosis is acceptable
2. Never received TACE/ chemotherapy/ radiotherapy or targeted agents prior to this study.
3. Patients should be either in BCLC clinical stage B (multinodular asymptomatic tumors without extra-hepatic spread or portal vein invasion) with or without unilateral secondary or tertiary branches of portal vein invasion. Main portal vein invasion or extra-hepatic spread is not allowed.
4. Child-Pugh functional class A or B.
5. Measurable disease using mRECIST criteria. At least 1 measurable lesion must be present.
6. ECOG performance status 0 to 1.
7. Age > 18 years
8. Both men and women enrolled in this trial must use adequate birth control measures during the course of the trial and 4 weeks after the completion of trial
9. Informed consent must be obtained prior to study initiation.
10. Total bilirubin < 3.0 mg/dL with no evidence of biliary tract obstruction.
11. Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5 × upper limit of normal.
12. Absolute neutrophil count > 1000/mm3; Platelets ≧ 60x109/L.
13. Serum creatinine < 2 x ULN.
14. Antiviral treatment for hepatitis B or C is allowed except for interferon.

Exclusion Criteria:

1. BCLC stage A.
2. Presence of extrahepatic metastasis.
3. Child-Pugh score =C
4. Significant cardiac disease.
5. Serious bacteria infection requiring systemic antibiotics.
6. Pregnancy
7. Expected non-compliance.
8. Uncontrolled illness including, but not limited to, ongoing infection, congestive hear failure, unstable angina pectoris, cardiac arryhythmia, or psychiatric illness.
9. Bleeding esophageal or gastric varices within three months without ligation or sclerosis injection therapy.
10. Subjects with known HIV infection.
11. ECOG status > or = 2

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-08; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Complete remission | 3 years

SECONDARY OUTCOMES:
Time to partial (including complete) response | 3 years
Time-to-tumor-progression (TTP) | 3 years
Progression free survival (PFS). | 3 years
Overall survival (OS) | 3 years
Safety and tolerability of TACE plus sorafenib therapy recorded and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Chau-Ting Yeh, MD/PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Result] Liang KH, Lin CL, Chen SF, Chiu CW, Yang PC, Chang ML, Lin CC, Sung KF, Yeh C, Hung CF, Chien RN, Yeh CT. GALNT14 genotype effectively predicts the therapeutic response in unresectable hepatocellular carcinoma treated with transcatheter arterial chemoembolization. Pharmacogenomics. 2016 Mar;17(4):353-66. doi: 10.2217/pgs.15.179. Epub 2016 Feb 12. PMID 26871639
- [Derived] Chen WT, Lin SM, Lee WC, Wu TJ, Lin CC, Shen CH, Chang ML, Lin CL, Yeh CT. GALNT14 genotype-guided chemoembolization plus sorafenib therapy in hepatocellular carcinoma: a randomized trial. Hepatol Int. 2022 Feb;16(1):148-158. doi: 10.1007/s12072-021-10283-7. Epub 2022 Jan 4. PMID 34982369